CLINICAL TRIAL: NCT00966537
Title: The 3-Dimensional Ultrasound for Fetal Anomaly Scan.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Liat Gindes, Sheba Medical Center
Other Study IDs: SHEBA-09-4936-LG-CTIL
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Pregnancy
Keywords: to study the clinical application of 3D/4D ultrasound for fetal scanning; to study the clinical application of 3D/4D ultrasound for pelvic scanning;; to demonstrate how to optimally display the different organs.; to correlate our findings with other diagnostic tools like MRI, CT;; to correlate our findings with clinical outcome.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is 1) to study the clinical application of 3D/4D ultrasound for fetal scanning during pregnancy; 2) ) to study the clinical application of 3D/4D ultrasound for pelvic scanning; 3) to demonstrate how to optimally display the different organs. 4) to correlate our findings with other diagnostic tools like MRI, CT; 5) to correlate our findings with clinical outcome.

DETAILED DESCRIPTION:
A prospective studies of patients that coming to the ultrasound (US) unit in Sheba Medical Center from November 2007 for diagnostic US examination.

Patients will receive information of the study (printed and oral) and will ask to sign informed consent to act as a research subject and permission to use personal heath information for research.

Studies is performed using commercially available ultrasound equipment (Voluson 730 Expert, General Electric Healthcare, Kretztechnik, Zipf, Austria) with volumetric abdominal RAB 4-8 MHz and volumetric transvaginal RIC 5-9 MHz transducer probes.

During the examination of the patient pictures and 3D/4D volumes will acquired either by static 3D or 4D Volume or STIC (Spacio Temporal Image Corelation), Contrast Imaging in plane C (VCI-C) with and without Doppler (Color, Power and High Definition) and with B-flow. Image quality will be assessed in various modes. For optimizing the image volumes manipulations will be performed by positioning of the

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman who come for fetal anomaly scan.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant woman
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel